CLINICAL TRIAL: NCT05462405
Title: Microneurography MSNA Measurements for Evaluating the Effect of BackBeat Medical Cardiac Neuromodulation Therapy (CNT) on Sympathetic Activity: An Acute Study
Brief Title: Evaluation of Sympathetic Activity Effects by the BackBeat Medical Cardiac Neuromodulation Therapy (CNT).
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: BackBeat Medical Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CS-09 BBM MSNA
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Hypertension
Keywords: Moderato implant
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Indirect evidence [see reference 1] shows that CNT may decrease the level of sympathetic activity locally (in the heart) and systemically. However, this effect was never directly measured in an experiment. It is also theorized that the decrease of sympathetic activity may persist for some time after CNT delivery is stopped, but this has to be verified using direct sympathetic activity level measurement. Such direct evidence of sympathetic activity reduction may enable application of CNT therapy to other diseases and patients that do not have adequate therapies today, such as heart failure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): All subjects enrolled will be in the same experimental group.
  Interventions: Procedure: Experimental group

INTERVENTIONS:
Procedure: Experimental group — In the setting phase subjects will be in recumbent position. A microneurography needle (0.2mm diameter isolated Tungsten micro-electrode) will be placed under the skin. An identical (not isolated) reference needle tip will be inserted within 2 cm of the first electrode. These are connected to a recording system (ADInstruments PowerLab). Once sympathetic activity can be measured using the needles, a sympathetic specific test will be used to calibrate the measurement and recording system. In the testing phase sequential pacing and CNT delivery will be programmed for a few minutes, the whole procedure expected to last less than 2 hours.

SUMMARY:
Measurement and recording of Muscle Sympathetic Neural Activity (MSNA) using microneurography, will be applied to subjects who have been already implanted with a Moderato IPG delivering the BackBeat CNT and/or pacing signals. Several tests will be performed by experienced professionals to ensure the acquired sympathetic nerve signals arise from the targeted nerve source.

The Moderato Programmer will be then used to program different sets of CNT for several minutes with a several minutes interval between delivery periods. This delivery pattern is used will allow to acquire sympathetic nerve signals with and without CNT. Subject blood pressure, respiration and ECG data will be collected and recorded, both for safety and for evaluation of CNT dependent secondary indicators of sympathetic activity.

DETAILED DESCRIPTION:
This will be a multi-center , open-label, non-randomized acute pilot study. The Moderato System is approved for marketing in Europe (has a CE mark) for standard pacing and the treatment of high blood pressure in patients requiring standard cardiac pacing. The therapy delivered by the Moderato system is referred to as CNT (Cardiac Neuromodulation Therapy).

Measurement and recording of Muscle Sympathetic Neural Activity (MSNA) using microneurography, has been used extensively [see reference 4,5]. A small, thin metal needle is inserted through the skin near the knee in proximity to a major nerve that is close to the skin (a few millimeters depth). The electrical activity of the nerve measured by the needle is a direct indication of peripheral sympathetic activity.

This measurement technique will be applied to subjects who are already implanted with a Moderato IPG that can deliver the BackBeat CNT pacing signals, whether CNT pacing was activated or not.

In recumbent position (lying in a bed), insertion of a microneurography needle (FHC 35mm long, 0.2mm diameter Tungsten microelectrodes model UNP35F2U) to the correct recording position is attempted for no more than 1 hour. This has been successful in approximately 75% of patients in previous MSNA studies. An identical reference needle is inserted within 2 cm of the first electrode. The needles are connected to a recording system (ADInstruments PowerLab). Once sympathetic activity can be measured using the needles, a cold pressor test is performed. In this test, the subject's hand is placed in cold water for up to 2 minutes. This test is known to affect sympathetic activity and is used to calibrate the measurement and recording system.

The Moderato Programmer is then used to program the implanted Moderato IPG to deliver different sets of CNT pacing signals parameters, each for several minutes with a several minutes interval between delivery periods. This delivery pattern is used in order to measure the effect of CNT pacing signals delivery on sympathetic activity level both during and after CNT pacing signals delivery. Subject blood pressure, respiration and ECG data is also collected and recorded, both for safety reasons and to evaluate the effect of CNT on secondary indicators of sympathetic activity.

After the different CNT pacing signal sets are delivered, the microneurography needles will be removed, the patient disconnected from all other measurement devices, and the procedure concluded.

Patients will be considered as having completed the study at the conclusion of the acute procedure unless a safety event is observed during the acute procedure in which case the patients will be followed until the event has been resolved.

ELIGIBILITY:
Inclusion Criteria:

* Subject is already implanted with a Moderato IPG that can be used to deliver CNT pacing signals, whether CNT pacing was activated or not.
* Subject is willing and able to comply with the study and procedures.

Exclusion Criteria:

* Subject is dependent on 100% ventricular pacing.
* Subject has symptoms of heart failure, NYHA Class III or greater.
* Subject has an ejection fraction of 25% or less
* Subject's systolic blood pressure is less than 100 mm Hg on the day of recording.
* Subject has decompensated heart failure
* Subject has significant (>3+) mitral regurgitation, aortic regurgitation, or aortic stenosis
* Subject has permanent atrial fibrillation.
* Subject has Atrial fibrillation on the day of the study.
* Subject has hypertrophic cardiomyopathy, restrictive cardiomyopathy, or interventricular septal thickness ≥15 mm.
* Subject is on dialysis
* Subject has prior neurological events (stroke or TIA) within the past year or a neurological event (stroke) at any prior time that has resulted in residual neurologic deficit.
* Subject has a history of autonomic dysfunction.
* Women who are pregnant or breast-feeding.
* Subject cannot or is unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-12-10 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Sympathetic activity will be calculated as burst frequency (bursts/min) and as burst incidence (bursts/100 heartbeats). A change in the nerve activity occurring between pacing and CNT is expected. | through study completion (18 months)
  Nerve firing is organised in burst activity which can be detected by the data acquisition system

SECONDARY OUTCOMES:
A change in Systolic Blood Pressure | through study completion (18 months)
  CNT main action is a reduction of the Systolic Blood Pressure

CONTACTS AND LOCATIONS:
Overall Officials: Bela Merkely, D, Ph.D., Principal Investigator — Heart and vascular Centre, Semmelweiss University
Locations (1):
- Semmelweis University Heart and Vascular Center, Budapest, Hungary

REFERENCES:
- [Result] Heusser K, Tank J, Engeli S, Diedrich A, Menne J, Eckert S, Peters T, Sweep FC, Haller H, Pichlmaier AM, Luft FC, Jordan J. Carotid baroreceptor stimulation, sympathetic activity, baroreflex function, and blood pressure in hypertensive patients. Hypertension. 2010 Mar;55(3):619-26. doi: 10.1161/HYPERTENSIONAHA.109.140665. Epub 2010 Jan 25. PMID 20101001
- [Result] Georgakopoulos D, Little WC, Abraham WT, Weaver FA, Zile MR. Chronic baroreflex activation: a potential therapeutic approach to heart failure with preserved ejection fraction. J Card Fail. 2011 Feb;17(2):167-78. doi: 10.1016/j.cardfail.2010.09.004. Epub 2010 Oct 29. PMID 21300307
- [Result] Hering D, Lambert EA, Marusic P, Walton AS, Krum H, Lambert GW, Esler MD, Schlaich MP. Substantial reduction in single sympathetic nerve firing after renal denervation in patients with resistant hypertension. Hypertension. 2013 Feb;61(2):457-64. doi: 10.1161/HYPERTENSIONAHA.111.00194. Epub 2012 Nov 19. PMID 23172929